CLINICAL TRIAL: NCT00764361
Title: A Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of NanoDOX™ Hydrogel(1.0% Doxycycline Monohydrate)in Diabetic Adult Subjects With Lower Extremity Ulcers Compared to Placebo Hydrogel.
Brief Title: Safety Study of Topical Doxycycline Gel for Adult Diabetic Lower Extremity Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanoSHIFT LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-DOX-NT/003
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic; Ulcer; Wound
MeSH Terms: conditions — Diabetic Foot; Ulcer; Wounds and Injuries | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NanoDOX™ Hydrogel (Experimental): 1.0% doxycycline gel
  Interventions: Drug: doxycycline
- Placebo (Placebo Comparator): placebo gel
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: doxycycline — 1.0% doxycycline gel applied topically to the wound once daily for 20 weeks
  Arms: NanoDOX™ Hydrogel
Drug: placebo gel — placebo gel applied topically to the wound once daily for 20 weeks
  Other Names: doxycycline
  Arms: Placebo

SUMMARY:
This study is a double-blind, one center, two-arm study with a two (2) week Run-In, evaluating the efficacy of a once-daily administration of NanoDOX™ Hydrogel topically applied to diabetic ulcers in concert with professionally administered Standard of Care (SOC) procedures as described by Standard Operating Procedure(s) of the Department of Veterans Administration Hospitals. During the run-in period patients with infected wounds will receive oral antibiotic and not be included in the topical portion of the study until the infection is shown by wound fluid analysis to be resolved. Following a two (2) week Run-In of all patients to receive SOC treatment for diabetic ulcers, patients would have either the investigational material or the placebo hydrogel applied as a part of their wound care. Each patient would receive 1.5 gm packets of either the test article or the placebo hydrogel for a once-daily home treatment accompanied by a dressing change.

DETAILED DESCRIPTION:
Study of NanoDOX vs placebo on diabetic ulcers of the lower leg/foot.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented history of type I or type II diabetes mellitus as defined by the American Diabetes Association
* Women of childbearing potential must have a negative urine pregnancy test at screening and at baseline, and:

  • Agree to use a double-barrier method of contraception during their participation in this study;
  * condoms (with spermicide) and hormonal contraceptives OR
  * condoms (with spermicide) and intrauterine device OR
  * intrauterine device and hormonal contraceptives OR
  * Abstains from sexual intercourse during their participation in this study OR
  * Is with a same-sex partner and does not participate in bisexual activities where there is a risk of becoming pregnant
* Have an ulcer on the lower extremity (distal to a line connecting the medial and lateral malleoli) that has been present for at least 3 weeks and that is 1.2 cm2 to 4.0 cm2 at initial screening
* Be able to apply study drug to their ulcer, or have a caregiver do it
* Adequate blood flow to target ulcer extremity as measured by transcutaneous oxygen tension (TcpO2) of >30mmHg
* Target ulcer is Grade I according to the Wagner Grading Scale
* Quantitative bacterial count of of < 1.0 x 1.0E5 per gram of tissue for non-infected ulcers
* Quantitative bacterial count of ≥ 1.0 x 1.0E5 per gram of tissue for infected ulcers

Exclusion Criteria:

* Be a pregnant or lactating woman or a female of childbearing potential who is not practicing acceptable form of birth control.
* Allergy to tetracycline, minocycline, demeclocycline, or any other known tetracycline derivative
* Have more than three chronic ulcers present at baseline
* Have undergone treatment with system corticosteroid or immunosuppressive therapy in the past 2 months
* Have connective tissue disease
* Currently be going through kidney dialysis for renal failure
* Have undergone treatment with doxycycline, Procuren®, or Regranex® within the last 30 days
* Have participated in another clinical research trial within the last 30 days
* Have a known history of osteomyelitis affecting to the area where the target ulcer is present
* Have any other concomitant condition which, in the opinion of the investigator, would make the subject unsuitable for the study.
* Subject has ulcers resulting from any cause other than diabetes (electrical burn, arterial insufficiency, chemical or radiation insult)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Abernethy, MD, Study Director — Alachua Government Services, Inc.
Locations (1):
- North Florida / South Georgia Veterans Administration Hospital, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited through the local veterans administration clinics
Pre-assignment Details: adult subjects with diabetic lower extremity ulcers were enrolled into the study after determination that the wound was not infected
Period: Overall Study
Arm/Group | NanoDOX™ Hydrogel | Placebo
Started | 8 | 7
Completed | 6 | 3
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NanoDOX™ Hydrogel | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.99 (11.53) | 68.86 (9.75) | 66.33 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Adverse Events
Description: Participants were monitored for 20 weeks during the study.
Time Frame: every 2 weeks
Measure: Number; unit: participants
Groups:
- NanoDOX™ Hydrogel: 1.0% doxycycline monohydrate gel
Arm/Group | NanoDOX™ Hydrogel | Placebo
Number analyzed (Participants) | 8 | 7
participants | 8 | 7

2. Secondary Outcome: Analyze the Molecular Changes in Pro-inflammatory Cytokine Levels That Occur in Diabetic Foot Ulcers as a Function of Healing Rate in the Presence /Absence of NanoDOX Hydrogel (1% Doxycycline Monohydrate Gel)
Time Frame: baseline, week 4, week 10, week 20
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | NanoDOX™ Hydrogel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
enrollment stopped before reaching the initial 40 subjects anticipated due to slow enrollment of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less